CLINICAL TRIAL: NCT06158763
Title: Development and Evaluation of a CBT-based Transdiagnostic Transcultural Web App for Mental Health Problems in Low and Middle-income Countries.
Brief Title: Development and Evaluation of a CBT-based Transdiagnostic Transcultural Web App for Mental Health Problems
Acronym: WCBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Association of Cognitive Therapists (Other)
Collaborators: World Psychiatric Association (WPA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PACTwCBT
Record Dates: First submitted 2023-09-01; First posted 2023-12-06 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Depression; Anxiety
Keywords: CBT; web application; depression; anxiety; self-help manual
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial to evaluate the feasibility and acceptability of delivering a new intervention. Participants who meet the inclusion criteria will be randomly allocated to intervention or control groups in a 1:1 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In the experimental group, a web-based application intervention will be provided.
  Interventions: Behavioral: Web-based CBT guided self-help Interventions
- Control Group (No Intervention): In the control group, the patients screened for depression or anxiety received treatment as usual (TAU). TAU consisted of standard care under the responsible family physician. TAU in low-income countries largely consists of pharmacological treatment with anti-depressant medication and follow-up in an outpatient clinic.

INTERVENTIONS:
Behavioral: Web-based CBT guided self-help Interventions — An existing CBT-based transdiagnostic self-help manual (Naeem et al., 2014) that has been used successfully in RCTs (Amin et al., 2020; Naeem et al., 2014) and has been used as an online intervention (http://khushiorkhatoon.com/) will be further adapted. The intervention consists of seven modules, including cognitive restructuring, problem-solving and behavioural activation.
  Arms: Experimental Group

SUMMARY:
This study aims to (1) develop a CBT-based transcultural, transdiagnostic interactive web app and (2) assess the feasibility, acceptability, and preliminary efficacy of this intervention.

DETAILED DESCRIPTION:
Three-quarters of the global burden of mental disorders, including depression and anxiety, lies in low and middle-income countries (LMICs) (WHO, 2017). However, the treatment gap for common mental disorders in LMICs is significant, with an estimated 90% of people in these settings unable to access appropriate mental health care (Vos et al., 2015).

Despite the strong evidence supporting effectiveness in several disorders, cognitive behaviour therapy (CBT) remains underutilized internationally due to the limited availability of comprehensive training programmes and qualified CBT-trained staff. (Myhr & Payne, 2006). However, self-help and GSH can be delivered online and have been found to be effective and feasible for individuals with depression and anxiety (Andrews et al., 2018). Furthermore, leveraging the unprecedented increase in cell phone users and internet technologies, as well as the decline in prices of handheld mobile devices, may overcome barriers to care and address the substantial mental health treatment gap in these settings (Lambert & Littlefield, 2009; Lewis et al., 2012; UN Foundation-Vodafone Foundation Partnership, 2020; WHO, 2011). We, therefore, propose the development and evaluation of a CBT-based transcultural, transdiagnostic interactive web app to address symptoms of depression, anxiety and stress.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 65 years
* At least 5 years of education
* Computer literate
* Owning a smartphone or a personal computer with a reliable internet connection
* Score of 8 or higher on Hospital Anxiety and Depression Scale-Depression or Anxiety scales as measured by their primary care clinician.

Exclusion Criteria:

* Substance use disorder according to DSM-5 criteria
* Significant cognitive impairment (for example, profound learning disability or dementia)
* Active psychosis as determined by their primary care clinician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of CBT-based transcultural, transdiagnostic interactive web app will be assessed | 12 weeks
  Feasibility \will be assessed through trial procedure, recruitment, retention and informal feedback from participants.
Acceptability of CBT-based transcultural, transdiagnostic interactive web app will be assessed | 12 weeks
  Acceptability will be assessed through trial procedure, recruitment, retention and informal feedback from participants.

SECONDARY OUTCOMES:
Clinical Measures | 12 weeks
  The Hospital Anxiety and Depression Scale (HADS) will be used to measure Anxiety and Depression. The HADS is a rating scale consisting of 14 items, Each of the items is scored on a 4-point Likert scale from 0 (not present) to 3 (considerable). The sum of the individual items provides subscale scores on the HADS-D and the HADS-A, which may range between 0 and 21. A cut-off point of ≥8 for each of the constituent subscales is used to indicate probable caseness.
The WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | 12 weeks
  The WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) will measure the functioning and disability. It covers 6 Domains, the scores assigned to each of the items - "none" (0), "mild" (1) "moderate" (2), "severe" (3) and "extreme" (4) - are summed.

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Association of Cognitive Therapists, Lahore, Punjab Province, Pakistan